CLINICAL TRIAL: NCT02079740
Title: An Open Label, Two-Part, Phase Ib/II Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of the MEK Inhibitor Trametinib and the BCL2-Family Inhibitor Navitoclax (ABT-263) in Combination in Subjects With KRAS or NRAS Mutation-Positive Advanced Solid Tumors
Brief Title: Trametinib and Navitoclax in Treating Patients With Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00461; NCI-2014-00461 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13-505; 9525 (Other: Dana-Farber Cancer Institute); 9525 (Other: CTEP); P30CA006516 (NIH); P50CA127003 (NIH); U01CA062490 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2025-01-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm; Unresectable Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; navitoclax; trametinib; omipalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (trametinib, navitoclax) (Experimental): Patients receive trametinib PO QD and navitoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. If unacceptable toxicity is observed, patients may receive trametinib PO QD on days 1-14.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Navitoclax; Procedure: Positron Emission Tomography; Drug: Trametinib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo conventional CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Navitoclax — Given PO
  Other Names: A-855071.0; ABT-263; BcI-2 Family Protein Inhibitor ABT-263
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Trametinib — Given PO
  Other Names: GSK 1120212; GSK 212; GSK-1120212; GSK-212; GSK1120212; GSK212; JTP 74057; JTP-74057; JTP74057; MEK Inhibitor GSK1120212

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of trametinib and navitoclax and how well they work in treating patients with solid tumors that have spread to other places in the body (advanced or metastatic). Trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Navitoclax inhibits members of the BCL2 family of proteins that are believed to play key roles in promoting the survival of cancer cells. It may stop the growth of cancer cells by blocking Bcl-2, Bcl-XL, and Bcl-w, proteins needed for cancer cell survival. Giving trametinib and navitoclax may help stop the growth of tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose-limiting toxicities of trametinib in combination with navitoclax, and the maximal doses at which both drugs can be safely administered together. (Phase Ib) II. To determine the response rate of the combination of trametinib and navitoclax in subjects with KRAS or NRAS mutation-positive advanced or metastatic solid tumors in disease-specific expansion cohorts. (Phase II) III. To confirm the safety and tolerability of trametinib and navitoclax in combination at the recommended phase 2 dose (RP2D) determined in the Phase 1b portion. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics of both drugs administered together. (Phase Ib) II. To assess for evidence of response to therapy. (Phase Ib) III. To evaluate the pharmacodynamic response to therapy in tumor biopsies. (Phase Ib) IV. To evaluate the pharmacodynamic response to therapy in tumor biopsies (first 15 patients enrolled overall). (Phase II)

OUTLINE: This is a phase Ib, dose-escalation study followed by a phase II study.

Patients receive trametinib orally (PO) once daily (QD) and navitoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. If unacceptable toxicity is observed, patients may receive trametinib PO QD on days 1-14. Patients also undergo computed tomography (CT), positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI) every 8 weeks following cycle 1 day 1, biopsy on day 15 or 22 of cycle 1, and collection of blood samples on day 1 of cycles 2, 4, 8, and 12.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically- or cytologically-confirmed diagnosis of KRAS or NRAS mutation-positive malignancy that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective; patients must have activating mutations affecting codons 12, 13, 61, or 146 as determined in a Clinical Laboratory Improvement Amendments (CLIA)-certified lab to be eligible for this study
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm by chest x-ray or as >= 10 mm with CT scan, MRI, or calipers by clinical exam
* Participants must have received at least one line of prior systemic chemotherapy and must have experienced documented radiographic progression or intolerance on this therapy
* Paired pre-treatment and post-treatment biopsies are required for all patients on Part 1 and first 15 patients in Part 2; participants must have available archival tumor tissue (at least 20 unstained slides); if archival tissue is not available or is found not to contain tumor tissue, a fresh biopsy is required; if a patient is having a tumor biopsy, less than 20 unstained slides are acceptable with approval of the principal investigator (PI); biopsies will only be performed in a given patient if they are not deemed to involve unacceptable risk based on the sites of disease and other concurrent medical conditions
* Age >= 18 years

  * Because no dosing or adverse event data are currently available on the use of trametinib in combination with navitoclax in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy of greater than 3 months
* Able to swallow and retain orally-administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events version 4 (CTCAE v 4) grade =< 1 (except alopecia) at the time of enrollment; this requirement to return to =< grade 1 does not apply to immune checkpoint inhibitor related endocrinopathies (e.g. thyroiditis, hypophysitis, etc.) that necessitate hormone replacement therapy including, but not limited to levothyroxine, cortisol, and testosterone; CTCAE v5.0 will be utilized beginning April 1, 2018
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,200/mcL (subjects may be treated with hematopoietic growth factors to achieve or maintain this level)
* Hemoglobin >= 9 g/dL
* Platelets >= 100 x 10^9/L
* Albumin >= 2.5 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (patients with Gilbert's syndrome may have serum bilirubin > 1.5 x ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.2 x institutional ULN
* Left ventricular ejection fraction >= institutional lower limit of normal (LLN) by echocardiogram (ECHO) or multi gated acquisition scan (MUGA)
* The effects of trametinib and navitoclax on the developing human fetus are unknown. For this reason, women of child-bearing potential and men with a female partner of child bearing potential must agree to use adequate contraception using one of the methods listed below prior to study entry, for the duration of study participation, and up to 4 months following completion of therapy

  * Total abstinence from sexual intercourse (minimum one complete menstrual cycle prior to study drug administration)
  * Vasectomized male subject or vasectomized partner of female subjects
  * Hormonal contraceptives (oral, parenteral, transdermal or vaginal ring) for at least 3 months prior to study drug administration; if the subject is currently using a hormonal contraceptive, she should also use a barrier method during this study and for 1 month after study completion
  * Intrauterine device (IUD)
  * Double-barrier method: male condom plus diaphragm or vaginal cap with spermicide (contraceptive sponge, jellies or creams)
  * Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception; additionally, male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the study and for 4 months following completion of therapy
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to initiation of treatment; women will be considered not of childbearing potential if they are surgically sterile (bilateral oophorectomy or hysterectomy) and/or post-menopausal (amenorrheic for at least 12 months); should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; the potential hazard to the fetus should be explained to the patient and partner (as applicable)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of another malignancy; exception: patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer or any carcinoma in situ and/or patients with indolent second malignancies, are eligible; consult the Cancer Therapy Evaluation Program (CTEP) medical monitor if unsure whether second malignancies meet the requirements specified above
* History of interstitial lung disease or pneumonitis
* Any major surgery, extensive radiotherapy (> 15 days of treatment), chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to first dose of study treatment and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to first dose of study treatment
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of study drug(s) and during the study
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; exception: patients with brain metastases will be allowed on study if they have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of central nervous system (CNS) disease progression as determined by CT or MRI within 21 days prior to the first dose of study drug
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to trametinib, or excipients or to dimethyl sulfoxide (DMSO), or to compounds of similar chemical or biologic composition to navitoclax
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment; (note: megestrol [Megace] if used as an appetite stimulant is allowed)
  * Concurrent treatment with bisphosphonates is permitted; however, treatment must be initiated prior to the first dose of study therapy; prophylactic use of bisphosphonates in patients without bone disease is not permitted, except for the treatment of osteoporosis
  * Because the composition, pharmacokinetics (PK), and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
  * Due to the expected dose-limiting toxicity of thrombocytopenia, the following concomitant medications are not allowed during navitoclax administration: Warfarin, clopidogrel (plavix), ibuprofen, tirofiban (aggrastat), and other anticoagulants, drugs, or herbal supplements that affect platelet function are excluded, with the exception of low-dose anticoagulation medications (such as heparin) that are used to maintain the patency of a central intravenous catheter; aspirin will not be allowed within 7 days prior to the first dose of navitoclax or during navitoclax administration; however, subjects who have previously received aspirin therapy for thrombosis prevention may resume a low dose (i.e., maximum 100 mg QD) of aspirin if platelet counts are stable (>= 50,000/mm^3) through 6 weeks of navitoclax administration; all decisions regarding treatment with aspirin therapy will be determined by the investigator in conjunction with the medical monitor
* Preclinical studies indicate that navitoclax is metabolized by CYP3A4, is a moderate inhibitor of CYP2C8, and is a strong inhibitor of CYP2C9; therefore, caution should be exercised when dosing navitoclax concurrently with CYP2C8 and CYP2C9 substrates; common CYP2C8 substrates include paclitaxel, statins, and glitazones, whereas CYP2C9 substrates include phenytoin and warfarin; when possible, investigators should switch to alternative medications or monitor the patients closely (particularly in the case of medications that have a narrow therapeutic window such as warfarin; use of warfarin is specifically prohibited while on study); CYP3A inhibitors such as ketoconazole and clarithromycin are not allowed 7 days prior to the first dose of navitoclax or during navitoclax administration

  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
  * Patient instructions and information of possible drug interactions will be given to all patients upon enrollment in this study
* History or current evidence/risk of retinal vein occlusion (RVO)
* History or evidence of cardiovascular risk including any of the following:

  * Left ventricle ejection fraction (LVEF) < LLN
  * A QT interval corrected for heart rate using the Bazett's formula QTcB >= 480 msec
  * History or evidence of current clinically significant uncontrolled arrhythmias (exception: patients with controlled atrial fibrillation for > 30 days prior to enrollment are eligible)
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to randomization
  * History or evidence of current >= class II congestive heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * Treatment-refractory hypertension defined as a blood pressure of systolic > 140 mmHg and/or diastolic > 90 mmHg which cannot be controlled by anti-hypertensive therapy
  * Known cardiac metastases
  * Patients with intra-cardiac defibrillators
* Known hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (patients with chronic or cleared HBV and HCV infection are eligible); patients with human immunodeficiency virus (HIV) are not eligible if on anti-retroviral medications
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Subject has an underlying condition predisposing them to bleeding or currently exhibits signs of clinically significant bleeding
* Subject has a recent history of non-chemotherapy-induced thrombocytopenic-associated bleeding within 1 year prior to the first dose of study drug
* Subject has a significant history of cardiovascular disease (e.g., myocardial infarction [MI], thrombotic or thromboembolic event in the last 6 months)
* Pregnant women or nursing mothers; animal reproductive studies have not been conducted with trametinib or navitoclax; therefore, the study drug must not be administered to pregnant women or nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2026-03-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan B Corcoran, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg; Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg; Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg; Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg; Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg; Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg; Cohort 4C = Trametinib 2 mg + Navitoclax 200 mg; Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg; Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg: During Phase 1b dose escalation, participants received trametinib orally (PO) once daily (QD) and navitoclax PO QD on days 1-28 of each cycle until disease progression or unacceptable toxicity.
  A 7-day lead-in dosing of Navitoclax 150 mg will be evaluated in Cycle 1 for dose levels 3-7 before proceeding to their target doses:
  * Schedule A = 7-day lead-in dosing of navitoclax as a single agent, prior to the initiation of trametinib dosing.
  * Schedule B = 7-day lead-in dosing of navitoclax simultaneous with the initiation of trametinib dosing.
  Dose levels 1-3 will be enrolled according to Schedule A (i.e., cohorts 1A, 2A, 3A). If significant safety concerns are noted, study will proceed according to Schedule A (i.e., cohorts 4A, 5A, 6A, 7A). If no significant safety concerns are noted, and it is deemed safe to proceed, dosing will return to dose level 1 according to schedule B (i.e., cohort 1B), then proceed directly cohort 3B.
  If >1 DLT within cohort 1B or 3B, then Schedule B will be abandoned, and study will proceed with cohorts 4A, 5A, 6A, 7A. If cohort 3B is completed with </= 1 DLT, and Schedule B demonstrates a comparable or improved safety profile relative to Schedule A, then study will proceed with cohorts 4B, 5B, 6B, 7B.
  If, however, unacceptable toxicity is observed at a given dose level independent of Schedule A or B, then an alternative dosing Schedule C will be explored with Trametinib dosing on days 1-14 only, beginning at last dose level completed.
- Expansion Cohort 1 = Pancreatic Cancer; Expansion Cohort 2 = GYN Cancer; Expansion Cohort 3 = Lung Cancer; Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types: Phase 2 expansion cohorts use recommended phase 2 dosing (RP2D) determined in Phase 1b. Participants with KRAS or NRAS mutation-positive solid tumors will be enrolled into up to 4 different disease-specific expansion cohorts:
  1. Pancreatic Cancer
  2. GYN Cancer
  3. Lung Cancer
  4. all other NRAS mutation-positive solid tumor types exclusive of pancreatic, GYN, and lung cancers
  Initially 12 participants will be enrolled to each expansion cohort in Stage 1. If no responses are observed in a given cohort among the first 12 patients, then that cohort will be stopped for futility. However, if one or more responses are observed in a given cohort, the cohort will proceed to Stage 2, and an additional 13 patients will be enrolled for a total of 25 patients in that cohort.
Period: Phase 1b: Dose Escalation
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg | Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 4C = Trametinib 2 mg + Navitoclax 200 mg | Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg | Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg | Expansion Cohort 1 = Pancreatic Cancer | Expansion Cohort 2 = GYN Cancer | Expansion Cohort 3 = Lung Cancer | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types
Started | 3 | 3 | 3 | 3 | 8 | 3 | 3 | 8 | 4 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 6 | 4 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Concurrent anticoagulation prohibited on study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Phase 2: Expansion Cohorts
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg | Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 4C = Trametinib 2 mg + Navitoclax 200 mg | Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg | Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg | Expansion Cohort 1 = Pancreatic Cancer | Expansion Cohort 2 = GYN Cancer | Expansion Cohort 3 = Lung Cancer | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 25 | 7 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 25 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg | Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 4C = Trametinib 2 mg + Navitoclax 200 mg | Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg | Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg | Expansion Cohort 1 = Pancreatic Cancer | Expansion Cohort 2 = GYN Cancer | Expansion Cohort 3 = Lung Cancer | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 8 | 3 | 3 | 8 | 4 | 14 | 25 | 7 | 12 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 1 | 2 | 6 | 2 | 2 | 7 | 3 | 9 | 16 | 5 | 8 | 66
  >=65 years | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 5 | 9 | 2 | 4 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3 | 5 | 2 | 1 | 8 | 2 | 8 | 25 | 4 | 8 | 69
  Male | 2 | 2 | 2 | 0 | 3 | 1 | 2 | 0 | 2 | 6 | 0 | 3 | 4 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  White | 3 | 3 | 2 | 3 | 6 | 2 | 2 | 6 | 3 | 13 | 23 | 6 | 11 | 83
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 6
Cancer Type [Count of Participants; unit: Participants]
  Pancreatic Cancer | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 14 | 0 | 0 | 0 | 21
  Lung Cancer | 1 | 2 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 0 | 16
  GYN Cancer | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 4 | 1 | 0 | 25 | 0 | 0 | 32
  Colorectal Cancer | 2 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 4 | 14
  Esophageal Cancer | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Melanoma | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 6
  Cholangiocarcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Gastric Cancer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Thyroid Cancer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: (Phase 1b) Maximal Tolerated Dose of Trametinib and Navitoclax
Description: Dose escalation uses a 3+3 enrollment design per dose level. The occurrence of 1 dose limiting toxicity (DLT) will prompt expansion of a given dose level to 6 participants. The occurrence of 2 DLTs in a given dose level will indicate that the maximal tolerated dose (MTD) has been exceeded, and expansion of the prior dose level to 6 participants will occur, if not already performed. The recommended phase 2 dose (RP2D) will be the highest dose level at which no more than 1 out of 6 participants experiences a DLT. Dose escalation will proceed until the MTD/RP2D have been determined.
Time Frame: Within the first 42 days of treatment
Measure: Number; unit: milligrams per day
Groups:
- Treatment (Trametinib, Navitoclax): Patients receive trametinib PO QD and navitoclax PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. If unacceptable toxicity is observed, patients may receive trametinib PO QD on days 1-14.
  Biopsy: Undergo biopsy
  Biospecimen Collection: Undergo collection of blood samples
  Computed Tomography: Undergo conventional CT or PET/CT
  Magnetic Resonance Imaging: Undergo MRI
  Navitoclax: Given PO
  Positron Emission Tomography: Undergo PET/CT
  Trametinib: Given PO
Arm/Group | Treatment (Trametinib, Navitoclax)
Number analyzed (Participants) | 38
milligrams per day
  Trametinib on Days 1-14 | 2
  Navitoclax on Days 1-28 | 250

2. Primary Outcome: (Phase 1b) Dose-Limiting Toxicities of Trametinib and Navitoclox
Description: Dose-limiting toxicity (DLT) are adverse events (AEs) that are serious enough to prevent an increase in dose level of that treatment. Grading based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. CTCAE version 5.0 will be utilized beginning April 1, 2018.
Time Frame: Within the first 42 days of treatment
Population: In Cohort 3B, 2 of 8 participants were deemed not evaluable for DLT. In Cohort 5C, 2 of 8 participants were deemed not evaluable for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg | Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 4C = Trametinib 2 mg + Navitoclax 200 mg | Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg | Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 3 | 3 | 6 | 4
Participants
  Grade 3 AST/ALT increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 4 hypokalemia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Bilirubin increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Grade 3 Enterocolitis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: (Phase 2) Response Rate
Description: Response rate is defined as the number of participants who achieve complete response (CR) or partial response (PR), according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1:
  * CR = Disappearance of target lesion(s). Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  * PR = At least a 30% decrease in the sum of the longest diameter(s) of target lesion(s)
  Participants are considered evaluable for response if they had measurable disease present at baseline, received at least one cycle of therapy, and had their disease re-evaluated at least once after initiating therapy.
Time Frame: Up to 6 months
Population: There were a total of 10 participants in phase 2 that were not evaluable for response because they did not have a restaging scan-- 1 from expansion cohort 1, 6 from expansion cohort 2, 1 from expansion cohort 3, and 2 from expansion cohort 4.
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort 1 = Pancreatic Cancer | Expansion Cohort 2 = GYN Cancer | Expansion Cohort 3 = Lung Cancer | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types
Number analyzed (Participants) | 11 | 19 | 5 | 8
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 6 | 0 | 1

4. Primary Outcome: (Phase 2) Progression-free Survival
Description: Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progressive disease (PD) or death, whichever occurs first.
  PD is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1 as at least a 20% increase in the (sum of the) longest diameter(s) of target lesion(s), and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to 31 months
Measure: Mean (Full Range); unit: months
Arm/Group | Expansion Cohort 1 = Pancreatic Cancer | Expansion Cohort 2 = GYN Cancer | Expansion Cohort 3 = Lung Cancer | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types
Number analyzed (Participants) | 12 | 25 | 6 | 10
months | 1.37 [0.60 to 2.87] | 5.87 [0.37 to 31.60] | 6.57 [1.33 to 26.77] | 5.17 [0.03 to 30.97]

5. Primary Outcome: (Phase 2) Treatment Emergent Adverse Events
Description: Treatment emergent adverse events (TEAEs) are undesirable events not present prior to study treatment, or an already present event that worsens either in intensity or frequency while on treatment. TEAEs are assessed as grade 3 or higher according to Common Terminology Criteria for Adverse Events (CTCAE) criteria version 4.0. CTCAE criteria version 5.0 will be utilized beginning April 1, 2018. TEAEs are also assessed as possibly, probably, or definitely related to study treatment.
Time Frame: up to 29 months on treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Expansion Cohort 1 = Pancreatic Cancer | Expansion Cohort 2 = GYN Cancer | Expansion Cohort 3 = Lung Cancer | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types
Number analyzed (Participants) | 12 | 25 | 6 | 10
Participants
  Grade 3 abdominal pain | 1 | 0 | 0 | 0
  Grade 3 ALT increase | 0 | 3 | 1 | 0
  Grade 3 anemia | 1 | 1 | 0 | 1
  Grade 3 AST increase | 0 | 2 | 0 | 0
  Grade 3 blood bilirubin increased | 0 | 1 | 0 | 0
  Grade 3 dehydration | 0 | 1 | 0 | 0
  Grade 3 diarrhea | 0 | 1 | 0 | 0
  Grade 3 hypertension | 0 | 0 | 0 | 1
  Grade 3 hypokalemia | 0 | 0 | 1 | 0
  Grade 3 hyponatremia | 0 | 1 | 0 | 0
  Grade 3 neutrophil count decrease | 0 | 4 | 1 | 0
  Grade 4 neutrophil count decrease | 0 | 1 | 0 | 0
  Grade 3 platelet count decrease | 1 | 2 | 0 | 4
  Grade 3 white blood cell decrease | 0 | 3 | 0 | 0

6. Secondary Outcome: (Phase 1b) Pharmacokinetic Parameter Cmax for Trametinib and Navitoclax When Administered in Combination
Description: Pharmacokinetic blood draw samples collected for the following parameter and reported as mean values per day: maximum observed plasma drug concentration (Cmax).
  Schedule A:
  * C1 D7 = pre-nav (0h) then 2h, 4h, 6h, 8h
  * C1 D8 = pre-tram (-1h = 23h post-nav)
  * C1 D21 = pre-tram (-1h); pre-nav (0h); then 2h, 4h, 6h, 8h post-nav
  * C1 D22 = pre-tram (-1h = 23h post-nav)
  * D1 of Cycle 2,4,8,12 (single trough) = pre-tram (-1h)
  Schedule B:
  * C1 D7, D14 = pre-tram (-1h); pre-nav (0h); then 2h, 4h, 6h, 8h post-nav
  * C1 D8, D15 = pre-tram (-1h = 23h post-nav)
  * D1 of Cycle 2,4,8,12 (single trough) = pre-tram (-1h)
  Schedule C:
  * C1 D7, D14 = pre-navitoclax (0h) then 2h, 4h, 6h, 8h
  * C1 D8, D15 = pre-trametinib (-1h = 23h post-navitoclax)
  * D1 of Cycle 2,4,8,12 (single trough) = pre-nav (0h)
Time Frame: Cycle 1 day 7 and day 21
Population: No data was collected for this outcome for phase 1 cohorts 1B, 3B, 3C, 4C, 5C or 6C.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg
Number analyzed (Participants) | 3 | 3 | 2
ng/mL
  Day 7 Navitoclax Cmax | 3120.0 [1710.0 to 4190.0] | 2374.0 [562.0 to 4480.0] | 3040.0 [2890.0 to 3190.0]
  Day 21 Navitoclax Cmax | 2325.0 [374.0 to 4740.0] | 1349.0 [347.0 to 1860.0] | 1405.0 [1380.0 to 1430.0]
  Day 21 Trametinib Cmax | 12.2 [8.37 to 20.5] | 19.6 [14.2 to 29.8] | 23.2 [21.5 to 25.0]

7. Secondary Outcome: (Phase 1b) Pharmacokinetic Parameter AUC for Trametinib and Navitoclax When Administered in Combination
Description: Pharmacokinetic blood draw samples collected for the following parameter and reported as mean values per day: area under the concentration time curve from zero (pre-dose) to 24 hours (AUC 0-24).
  Schedule A:
  * C1 D7 = pre-nav (0h) then 2h, 4h, 6h, 8h
  * C1 D8 = pre-tram (-1h = 23h post-nav)
  * C1 D21 = pre-tram (-1h); pre-nav (0h); then 2h, 4h, 6h, 8h post-nav
  * C1 D22 = pre-tram (-1h = 23h post-nav)
  * D1 of Cycle 2,4,8,12 (single trough) = pre-tram (-1h)
  Schedule B:
  * C1 D7, D14 = pre-tram (-1h); pre-nav (0h); then 2h, 4h, 6h, 8h post-nav
  * C1 D8, D15 = pre-tram (-1h = 23h post-nav)
  * D1 of Cycle 2,4,8,12 (single trough) = pre-tram (-1h)
  Schedule C:
  * C1 D7, D14 = pre-navitoclax (0h) then 2h, 4h, 6h, 8h
  * C1 D8, D15 = pre-trametinib (-1h = 23h post-navitoclax)
  * D1 of Cycle 2,4,8,12 (single trough) = pre-nav (0h)
Time Frame: Cycle 1 day 7 and day 21
Population: No data was collected for this outcome for phase 1 cohorts 1B, 3B, 3C, 4C, 5C or 6C.
Measure: Mean (Full Range); unit: h*ng/mL
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg
Number analyzed (Participants) | 3 | 3 | 2
h*ng/mL
  Day 7 Navitoclax AUC | 52219.0 [26752.0 to 66795.0] | 35451.0 [9148.5 to 67610.0] | 48714.0 [48038.5 to 49390]
  Day 21 Navitoclax AUC | 30575.0 [7385.0 to 44056.0] | 24224.0 [6177.0 to 38322.0] | 25804.0 [24609.0 to 26999.0]
  Day 21 Trametinib AUC | 206.0 [160.0 to 308.0] | 311.0 [221.0 to 483.0] | 305.0 [283.0 to 329.0]

8. Secondary Outcome: (Phase 1b) Pharmacokinetic Parameter C0 for Trametinib and Navitoclax When Administered in Combination
Description: Pharmacokinetic blood draw samples collected for the following parameter and reported as mean values per day: trough plasma drug concentration (C0).
  Schedule A:
  * C1 D7 = pre-nav (0h) then 2h, 4h, 6h, 8h
  * C1 D8 = pre-tram (-1h = 23h post-nav)
  * C1 D21 = pre-tram (-1h); pre-nav (0h); then 2h, 4h, 6h, 8h post-nav
  * C1 D22 = pre-tram (-1h = 23h post-nav)
  * D1 of Cycle 2,4,8,12 (single trough) = pre-tram (-1h)
  Schedule B:
  * C1 D7, D14 = pre-tram (-1h); pre-nav (0h); then 2h, 4h, 6h, 8h post-nav
  * C1 D8, D15 = pre-tram (-1h = 23h post-nav)
  * D1 of Cycle 2,4,8,12 (single trough) = pre-tram (-1h)
  Schedule C:
  * C1 D7, D14 = pre-navitoclax (0h) then 2h, 4h, 6h, 8h
  * C1 D8, D15 = pre-trametinib (-1h = 23h post-navitoclax)
  * D1 of Cycle 2,4,8,12 (single trough) = pre-nav (0h)
Time Frame: Cycle 1 day 7 and day 21
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg
Number analyzed (Participants) | 3 | 3 | 2
ng/mL
  Day 7 Navitoclax C0 | 1156.7 [510 to 1520] | 1012.0 [314 to 1710] | 910.5 [551 to 1270]
  Day 21 Navitoclax C0 | 1110 [221 to 1860] | 584 [207 to 1080] | 949 [857 to 1040]
  Day 21 Trametinib C0 | 6.4 [4.8 to 9.43] | 9.7 [7.5 to 14.9] | 9.9 [8.8 to 11.1]

9. Secondary Outcome: (Phase 1b) Response Rate
Description: as for outcome 3
Time Frame: Up to 4 months
Population: There were a total of 6 participants in phase 1 that were not evaluable for response because they did not have a restaging scan-- 1 from cohort 1A (clinical progression), 3 from cohort 3B, and 2 from cohort 5C.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg | Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 4C = Trametinib 2 mg + Navitoclax 200 mg | Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg | Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 5 | 3 | 3 | 6 | 4
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

10. Secondary Outcome: (Phase 2) Pharmacokinetic Parameters for Trametinib and Navitoclax When Administered in Combination at Recommended Phase 2 Dose
Description: Pharmacokinetic (PK) blood draw samples collected for the following parameters:
  * Maximum observed plasma drug concentration (Cmax)
  * Area under the concentration time curve from zero (pre-dose) to 24 hours (AUC 0-24)
  * Pre-dose (trough) drug concentration at the end of the dosing interval (C0)
  * Half-life (t1/2)
  Recommended phase 2 dose (RP2D) schedule:
  - Day 1 of cycles 2, 4, 8, 12 = pre-trametinib (-1h)
Time Frame: Day 1 of cycles 2, 4, 8, and 12
Population: No data was collected for this outcome in the phase 2 expansion cohorts.
Arm/Group | Expansion Cohort 1 = Pancreatic Cancer | Expansion Cohort 2 = GYN Cancer | Expansion Cohort 3 = Lung Cancer | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: (Phase 1b and 2) Percent Change in Levels of Proteins/Messenger Ribonucleic Acids Implicated in Mitogen-activated Protein Kinase Signaling
Description: Paired pre-treatment and on treatment tumor biopsies will be obtained to assess the pharmacodynamic response to therapy (e.g., change in levels of proteins/mRNAs implicated in MAPK signaling). Results will be reported as a mean percent (%) change in MAPK transcripts day 15 vs day 0.
  Pre-treatment tumor tissue for analysis will be obtained either from archival tissue remaining from a participant's prior surgery, diagnostic biopsy, or other procedure performed during routine clinical care. Alternatively, study-related pre-treatment biopsies will be obtained between days -21 and -1 of treatment if necessary.
  On-treatment biopsies will be obtained after ~2 weeks of Cycle 1 combination dosing:
  * Phase 1b Schedule A = Day 22 +/- 7 days
  * Phase 1b Schedule B or C = Day 15 +/- 7 days
  * Phase 2 RP2D = Day 15 +/- 7 days
Time Frame: up to 50 days
Measure: Mean (Standard Error); unit: percentage of change MAPK transcripts
Groups:
- Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg; Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg; Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg; Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg; Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg; Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg; Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg; Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg: During Phase 1b dose escalation, participants received trametinib orally (PO) once daily (QD) and navitoclax PO QD on days 1-28 of each cycle until disease progression or unacceptable toxicity.
  A 7-day lead-in dosing of Navitoclax 150 mg will be evaluated in Cycle 1 for dose levels 3-7 before proceeding to their target doses:
  Schedule A = 7-day lead-in dosing of navitoclax as a single agent, prior to the initiation of trametinib dosing.
  Schedule B = 7-day lead-in dosing of navitoclax simultaneous with the initiation of trametinib dosing.
  Dose levels 1-3 will be enrolled according to Schedule A (i.e., cohorts 1A, 2A, 3A). If significant safety concerns are noted, study will proceed according to Schedule A (i.e., cohorts 4A, 5A, 6A, 7A). If no significant safety concerns are noted, and it is deemed safe to proceed, dosing will return to dose level 1 according to schedule B (i.e., cohort 1B), then proceed directly cohort 3B.
  If >1 DLT within cohort 1B or 3B, then Schedule B will be abandoned, and study will proceed with cohorts 4A, 5A, 6A, 7A. If cohort 3B is completed with </= 1 DLT, and Schedule B demonstrates a comparable or improved safety profile relative to Schedule A, then study will proceed with cohorts 4B, 5B, 6B, 7B.
  If, however, unacceptable toxicity is observed at a given dose level independent of Schedule A or B, then an alternative dosing Schedule C will be explored with Trametinib dosing on days 1-14 only, beginning at last dose level completed.
- Expansion Cohort 2 = GYN Cancer; Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types; Expansion Cohort 1 = Pancreatic Cancer: Phase 2 expansion cohorts use recommended phase 2 dosing (RP2D) determined in Phase 1b. Participants with KRAS or NRAS mutation-positive solid tumors will be enrolled into up to 4 different disease-specific expansion cohorts:
  Pancreatic Cancer GYN Cancer Lung Cancer all other NRAS mutation-positive solid tumor types exclusive of pancreatic, GYN, and lung cancers Initially 12 participants will be enrolled to each expansion cohort in Stage 1. If no responses are observed in a given cohort among the first 12 patients, then that cohort will be stopped for futility. However, if one or more responses are observed in a given cohort, the cohort will proceed to Stage 2, and an additional 13 patients will be enrolled for a total of 25 patients in that cohort.
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg | Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg | Expansion Cohort 2 = GYN Cancer | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types | Expansion Cohort 1 = Pancreatic Cancer
Number analyzed (Participants) | 1 | 1 | 2 | 1 | 4 | 2 | 2 | 1 | 6 | 1 | 2
percentage of change MAPK transcripts | 15.2 (0) | -98.3 (0) | -39.5 (25) | -98.3 (0) | 6.0 (67) | 8.7 (19) | -49.0 (50) | -42.5 (0) | 6.8 (99) | 132.0 (0) | 175.3 (229)

ADVERSE EVENTS:
Time Frame: Up to 34 months
Arm/Group | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg | Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg | Cohort 4C = Trametinib 2 mg + Navitoclax 200 mg | Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg | Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg | Expansion Cohort 1 = Pancreatic Cancer | Expansion Cohort 2 = GYN Cancer | Expansion Cohort 3 = Lung Cancer | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 2/3 | 3/3 | 7/8 | 3/3 | 3/3 | 6/8 | 3/4 | 10/12 | 14/25 | 4/6 | 6/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 1/3 | 1/8 | 0/3 | 1/3 | 0/8 | 1/4 | 1/12 | 2/25 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 8/8 | 3/3 | 3/3 | 7/8 | 4/4 | 11/12 | 22/25 | 5/6 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg (N=3) | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg (N=3) | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg (N=3) | Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg (N=3) | Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg (N=8) | Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg (N=3) | Cohort 4C = Trametinib 2 mg + Navitoclax 200 mg (N=3) | Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg (N=8) | Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg (N=4) | Expansion Cohort 1 = Pancreatic Cancer (N=12) | Expansion Cohort 2 = GYN Cancer (N=25) | Expansion Cohort 3 = Lung Cancer (N=6) | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A = Trametinib 1 mg + Navitoclax 150 mg (N=3) | Cohort 2A = Trametinib 1.5 mg + Navitoclax 150 mg (N=3) | Cohort 3A = Trametinib 1.5 mg + Navitoclax 200 mg (N=3) | Cohort 1B = Trametinib 1 mg + Navitoclax 150 mg (N=3) | Cohort 3B = Trametinib 1.5 mg + Navitoclax 200 mg (N=8) | Cohort 3C = Trametinib 1.5 mg + Navitoclax 200 mg (N=3) | Cohort 4C = Trametinib 2 mg + Navitoclax 200 mg (N=3) | Cohort 5C = Trametinib 2 mg + Navitoclax 250 mg (N=8) | Cohort 6C = Trametinib 2 mg + Navitoclax 300 mg (N=4) | Expansion Cohort 1 = Pancreatic Cancer (N=12) | Expansion Cohort 2 = GYN Cancer (N=25) | Expansion Cohort 3 = Lung Cancer (N=6) | Expansion Cohort 4 = All Other NRAS Mutation-positive Solid Tumor Types (N=10)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 6 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 3 | 2 | 5 | 21 | 3 | 6
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 3 | 12 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 3 | 1 | 2 | 1 | 1 | 3 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 7 | 4 | 7 | 18 | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 4 | 0 | 1
Blurred vision (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 3 | 3 | 2 | 6 | 1 | 3 | 6 | 3 | 5 | 17 | 3 | 5
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Edema face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Edema limbs (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 4 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Eye disorders other (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — stye
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 3 | 1 | 2 | 14 | 1 | 2
Fever (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 8 | 0 | 0
Floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital edema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
gastrointestinal disorders other specify (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — Hematochezia
gastrointestinal disorders other specify (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — Perifissural Bleeding With Bowel Movement
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
hepatobiliary disorders other specify (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — Hepatocellular Injury
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infections and infestations Other, specify (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — Oral Thrush
INR increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 2 | 7 | 2 | 0 | 4 | 1 | 1 | 13 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 2 | 4 | 13 | 2 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Periorbital edema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 2 | 2 | 3 | 3 | 5 | 0 | 2 | 6 | 1 | 10 | 18 | 3 | 5
PPE syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4 | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 2 | 3 | 1 | 1 | 5 | 3 | 3 | 16 | 1 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1 | 4 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3 | 0 | 5 | 1 | 1 | 4 | 1 | 1 | 10 | 1 | 5
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
White blood cell decreased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 9 | 1 | 1
Skin and subcutaneous tissue disorders Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — bleeding from tumor

LIMITATIONS AND CAVEATS:
The CRO (contract research organization) did not collect, measure, calculate, or report t1/2 (half-life) as part of their PK analysis. Therefore, the investigators do not have access to this information and cannot report it.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT02079740/Prot_SAP_001.pdf